CLINICAL TRIAL: NCT06794086
Title: SBRT Combined With PD-1 Monoclonal Antibody in Unresectable Colorectal Liver Metastases: A Prospective, Multicenter, Single-arm, Phase II Clinical Study (SPARKLE-L)
Brief Title: SBRT + PD-1 Monoclonal Antibody in Unresectable Colorectal Liver Metastases
Acronym: SPARKLE-L
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jun Huang (Other)
Responsible Party: Sponsor-Investigator, Jun Huang, Professor, Sixth Affiliated Hospital, Sun Yat-sen University
Organization: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2024366
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer; Liver Metastases
Keywords: Stereotactic body radiation therapy; PD-1 Monoclonal Antibody
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Radiosurgery; spartalizumab; sintilimab; Drug Therapy; Fluorouracil

STUDY DESIGN:
Intervention Model Description: SBRT plus PD-1 Monoclonal Antibody
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT plus PD-1 Monoclonal Antibody (Experimental): Enrolled patients will receive stereotactic body radiation therapy with a dose of 8-12 Gy in 5 fractions. Chemotherapy based on 5-FU combined with PD-1 monoclonal antibody immunotherapy will be administered before and after radiotherapy.
  Interventions: Radiation: Stereotactic body radiation therapy; Drug: PD-1 Monoclonal Antibody; Drug: Chemotherapy

INTERVENTIONS:
Radiation: Stereotactic body radiation therapy — Stereotactic body radiation therapy (SBRT) is a highly precise form of external beam radiation therapy used to treat tumors in various parts of the body. Enrolled patients will initiate SBRT treatment within 2 weeks after the first course of chemotherapy. Intensity-modulated radiation therapy (IMRT) will be used, with the gross tumor volume (GTV) receiving a dose of 8-12 Gy in 5 fractions, resulting in a total dose of 40-60 Gy. The biologically effective dose (BED) is equivalent to 72-132 Gy. The treatment will be administered from Monday to Friday.
Drug: PD-1 Monoclonal Antibody — PD-1 monoclonal antibody is a type of immunotherapy drug designed to treat various cancers by targeting the programmed death receptor-1 (PD-1) pathway.The PD-1 monoclonal antibody used in this study is sintilimab at a dose of 200 mg, administered via intravenous infusion on Day 1. Participants will be considered eligible only if they have completed four or more cycles of PD-1 monoclonal antibody treatment both before and after SBRT.
  Other Names: sintilimab
Drug: Chemotherapy — Chemotherapy regimens based on fluorouracil (5-FU), such as CAPOX with a 3-week cycle or mFOLFOX6/FOLFIRI/FOLFOXIRI with a 2-week cycle, may be combined with targeted therapy. During chemotherapy or chemoradiotherapy, optimal supportive care will be provided.
  Other Names: fluorouracil

SUMMARY:
To explore the efficacy and safety of stereotactic body radiation therapy (SBRT) combined with PD-1 monoclonal antibody in the treatment of unresectable colorectal cancer liver metastasis through a prospective study, providing high-level evidence-based medical evidence for the use of SBRT combined with PD-1 inhibitors in the treatment of unresectable colorectal cancer liver metastasis.

DETAILED DESCRIPTION:
For patients with unresectable colorectal cancer liver metastasis, this study aims to explore whether the combination of stereotactic body radiation therapy (SBRT) and PD-1 monoclonal antibody can improve the objective response rate (ORR), achieve better long-term survival benefits, and enhance quality of life. Additionally, the study will investigate the efficacy and safety of SBRT combined with PD-1 monoclonal antibody for treating liver metastases, with the goal of providing high-level evidence-based medical evidence for the use of local hypofractionated radiotherapy combined with PD-1 monoclonal antibody in the treatment of unresectable colorectal cancer liver metastasis.

This is a prospective, open-label, multicenter, single-arm, Phase II study. Patients with colorectal cancer will be eligible for enrollment if the hepatobiliary surgery team within the multidisciplinary team (MDT) deems the liver metastases unresectable, and the radiation oncology team within the MDT considers the liver metastases suitable for stereotactic body radiation therapy (SBRT).

Enrolled patients will receive hypofractionated radiotherapy with a dose of 8-12 Gy in 5 fractions. Chemotherapy based on 5-FU combined with immunotherapy will be administered before and after radiotherapy. Eight weeks (±2 weeks) after the completion of radiotherapy, radiological assessment or multi-site liver biopsy will be performed. The MDT will then decide on the subsequent management: maintenance chemotherapy or watch-and-wait (W&W) for patients achieving complete clinical response (cCR) or pathological complete response (pCR), or maintenance chemotherapy or discontinuation for patients who do not achieve cCR/pCR.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent, voluntarily signed and dated by the subject, must be obtained in accordance with regulatory and institutional guidelines before any procedures related to the study protocol that are not part of routine care are performed.
2. Patients with pMMR/MSS colorectal adenocarcinoma;
3. Age 18-75 years;
4. Patients with histologically or cytologically confirmed colorectal cancer liver metastasis, with or without extrahepatic oligometastatic lesions, who are deemed by the hepatobiliary surgeon within the multidisciplinary team (MDT) to be ineligible for upfront R0 resection of liver metastases (unresectability is defined as one or more of the following conditions: ① Involvement of both left and right branches of the portal vein at the first hepatic hilum; ② Involvement of ≥2 hepatic veins at the second hepatic hilum; ③ No indication for upfront R0 resection/ablation after MDT discussion);
5. Liver metastases are measurable by imaging (based on RECIST 1.1 criteria), with a maximum diameter of ≤6 cm;
6. Patients who have not previously received radiotherapy for liver metastases, or whose liver tissue near the planned irradiation site has not been previously irradiated, and who have at least 700 cc of liver volume outside the treatment area;
7. Previous hepatectomy, systemic chemotherapy, or local ablation therapy, or hepatic arterial infusion pump chemotherapy is allowed, with a washout period of 2 weeks;
8. Child-Pugh score Class A ;
9. ECOG performance status 0-1;
10. Peripheral blood counts and liver and renal function within allowable ranges (tested within 15 days before the start of treatment);
11. No history of other malignancies, not pregnant or breastfeeding, and effective contraception should be used during the study period and for 6 months after the last dose;
12. Life expectancy of ≥6 months.

Exclusion Criteria:

1. Active hepatitis, cirrhosis, or Child-Pugh score Class B or C;
2. Extrahepatic metastases: bone or brain metastases, or ≥3 unresectable lung metastases (according to the 8th edition of the UICC);
3. Unmeasurable liver metastases;
4. History of severe drug allergies (including allergies to platinum agents, 5-FU, LV, and 5-HT3 receptor antagonists);
5. Patients who have participated in or are currently participating in other clinical trials within the past 4 weeks;
6. History of prior treatment with anti-PD-1, PD-L1, PD-L2, CTLA-4, or any other specific T-cell costimulatory or checkpoint pathway-targeted therapies;
7. Severe electrolyte abnormalities;
8. Presence of gastrointestinal diseases, such as active gastric or duodenal ulcers, ulcerative colitis, or unresected tumors with active bleeding; or other conditions that may lead to gastrointestinal bleeding or perforation (Note: Gastrointestinal fistulas that have not healed after surgical treatment, such as rectovesical, rectourethral, or rectovaginal fistulas, are exclusionary unless a stoma has been created and there are no active symptoms);
9. History of arterial thrombosis or deep vein thrombosis within 6 months; history of bleeding or evidence of bleeding tendency within 2 months;
10. Pregnant or breastfeeding women, or women of childbearing potential with a positive pregnancy test before the first dose; or female participants unwilling to strictly practice contraception during the study, as well as their partners;
11. Patients with active autoimmune deficiency diseases requiring systemic treatment within the past 2 years (i.e., use of immunomodulators, corticosteroids, or immunosuppressive drugs);
12. Presence of other active malignancies (except for malignancies that have been treated with curative intent and have been disease-free for over 3 years, or in situ cancers that can be cured with adequate treatment);
13. Presence of severe ECG abnormalities or active coronary artery disease within 12 months before study entry, severe/unstable angina, newly diagnosed angina or myocardial infarction, or New York Heart Association (NYHA) Class II or higher congestive heart failure;
14. Patients with active infections (fever above 38°C due to infection);
15. Patients with poorly controlled hypercalcemia, hypertension, or diabetes;
16. Patients with severe pulmonary diseases (interstitial pneumonia, pulmonary fibrosis, severe emphysema, etc.);
17. Patients with psychiatric disorders affecting clinical management or a history of central nervous system diseases;
18. Patients with severe complications (intestinal obstruction, renal insufficiency, hepatic insufficiency, cerebrovascular disorders, etc.);
19. Presence of any CTCAE Grade 2 or higher toxicity from prior treatments that has not resolved (except for anemia, alopecia, and skin pigmentation);
20. Any unstable medical condition that may affect patient safety or compliance with the study;
21. Patients deemed by the investigator to be unsuitable for participation in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2027-01-20 (Estimated)

PRIMARY OUTCOMES:
ORR | 1 year
  Objective Response Rate

SECONDARY OUTCOMES:
DCR | 1 year
  Disease Control Rate
pCR | 1 year
  Pathological Complete Response
1 year PFS | 1 year
  Local Progression-Free Survival of 1 Year
1 year OS | 1 year
  Overall Survival of 1 Year
2 years PFS | 2 years
  Local Progression-Free Survival of 2 Years
2 years OS | 2 years
  Overall Survival of 2 Years
R0 resection rate | 1 year
  The Rate of Negative margins under microscopy
Acute toxicity reactions | 1 year
  Referring to the percentage of patients experiencing acute toxicities related to radiotherapy, chemotherapy, and immunotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Jun Huang, PhD., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China